CLINICAL TRIAL: NCT02807025
Title: Nasal, Tracheal and Bronchial Mucosal Lining Fluid(MLF) Sampling From Patients With Respiratory Diseases
Acronym: RESPI-SAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15/LO/0444
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-04

CONDITIONS: IPF; Sarcoidosis; Tuberculosis; Asthma; COPD; Healthy
MeSH Terms: conditions — Sarcoidosis; Tuberculosis; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Idiopathic Pulmonary Fibrosis(IPF): Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and Chronic Obstructive Pulmonary Disease (COPD). Similar sampling from healthy controls for comparative data.
- Sarcoidosis: Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and Chronic Obstructive Pulmonary Disease (COPD). Similar sampling from healthy controls for comparative data.
- Tuberculosis(TB): Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and Chronic Obstructive Pulmonary Disease (COPD). Similar sampling from healthy controls for comparative data.
- Chronic Obstructive Pulmonary Disease: Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and Chronic Obstructive Pulmonary Disease (COPD). Similar sampling from healthy controls for comparative data.
- Asthma: Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and Chronic Obstructive Pulmonary Disease (COPD). Similar sampling from healthy controls for comparative data.
- Healthy: Nasal, tracheal and bronchial sampling of MLF in patients from healthy controls for comparative data.

SUMMARY:
Nasal, tracheal and bronchial sampling of MLF in patients with idiopathic pulmonary fibrosis(IPF), sarcoidosis, tuberculosis(TB), asthma and COPD. Similar sampling from healthy controls for comparative data.

Aim: To characterise the molecular basis of the upper and lower airway mucosa inflammatory response in different respiratory diseases. To assess molecular biomarkers and signatures to see if these can aid diagnosis, stratification of these respiratory diseases. To direct personalised medicine and rationalise therapy.

Outcome measures:Measurement of levels of inflammation, coagulation, complement activation and fibrosis in MLF, transcriptomics from nasal curettage and airway brushings and to assess the tolerability of absorption procedures in these patients.

DETAILED DESCRIPTION:
Aim- To define the diagnosis, stratification and monitoring of IPF, sarcoidosis and TB, providing targets and biomarkers for new therapy. The investigators will study asthma and COPD patients with inflammation of the airways, and to compare with healthy control subjects. Characterising inflammation using upper airway sampling may eventually remove the requirement for invasive diagnostic bronchoscopy in these patients. The investigators shall assess the presence of cytokines, chemokines, together with complement, coagulation and fibrosis. The investigators propose to obtain opportunistic nasal, bronchial and tracheal mucosal samples from patients with IPF, sarcoidosis and TB. The investigators will compare these samples with healthy controls and with patients with asthma and COPD.

Objectives: Determining biomarkers and molecular signatures in terms of cytokines and chemokines, coagulation, complement activation and fibrosis in the MLF from the range of lung diseases Study design: This is a pilot study and the investigators shall obtain our study group from patients attending the bronchoscopy suite, specialist respiratory clinics and those being admitted to the wards at St Mary's Hospital under the Respiratory team. The investigators shall recruit patients with asthma and COPD,as well as age/ sex- matched healthy volunteers.

IPF, sarcoid and TB patients are usually undergoing bronchoscopy or endobronchial ultrasound(EBUS) and transbronchial needle aspiration(TBNA) for diagnostic purposes. Their diagnosis may only be confirmed after sampling is done after the bronchoscopy.

The patients included in the study will represent the following groups:

IPF at least 12 subjects Sarcoidosis at least 12 subjects TB at least 12 subjects COPD at least 12 subjects Asthma at least 12 subjects Healthy at least 12 subjects Study visits: Having identified patients suitable for this study, the study involves a single bronchoscopy, during which all airway sampling takes place. The investigators will recruit patients with asthma, COPD and healthy volunteers and they will be reimbursed for their participation, since bronchoscopy is not routinely part of their normal clinical care. They will be recruited by advertisements to the general public. They will be given relevant participant information sheet regarding this study by email or post.

Participants with confirmed or suspected IPF, sarcoidosis and TB who are due for a bronchoscopy will be identified during their routine clinical care and as part of their diagnostic work-up, and will not receive compensation.

ELIGIBILITY:
Inclusion criteria for all participants-

* Women of childbearing age should not be pregnant, planning to get pregnant or breastfeeding.
* Participants should have no upper respiratory tract infections in past 6 weeks.
* Participants should have no significant cardiovascular disease.
* Body mass index (BMI) should be between 18 and 39.
* Participants with signs or symptoms of significant nasal anatomical defects including hypertrophy of turbinates, major septum deviation, nasal polyposis or recurrent sinusitis and nasal mucosal defects, injury, ulceration will not undergo nasal sampling.
* All participants will have to be able to provide informed consent.

Inclusion Criteria:

* Healthy volunteer- no history of lung disease, age 18-65, BMI 18-39, PEF >90%, no reversibility, no atopy, non smoker/ ex smoker with >10PYH.
* Asthma- diagnosis of asthma, age 18-65, BMI 18-39, GINA mild, PEF >70%, reversibility with salbutamol or positive with histamine, well controlled on asthma questionnaire(ACQ <0.75), non smoker/ex smoker with <10PYH.
* IPF- HRCT suggestive ofILD/IPF, age 45-80, BMI 18-39, FVC >50%, DLCO 30-90%.
* Sarcoidosis- HRCT suggestive of sarcoidosis, age 18-95, BMI 18-39, FVC>50%, DLC0>30%.
* TB- same as sarcoidosis, including clinical history and/ or CT evidence of TB, age 18-65.
* COPD- diagnosis of COPD, age 45-65, age 18-39, gold stage 2, post bronchodilator FEV1 50-79%, FEV1/FVC ratio <70%,TLCO 60-80% or emphysema on HRCT,Smoker/ex smoker with >10PYH.

Exclusion Criteria:

* Healthy volunteer- use of anti-inflammatory meds including statins, antihistamines, NSAIDs, salicylates, anti-rheumatics, use of any OTC medications, URTI within the last six weeks, chronic inflammatory illness or CVS/ Resp disease/ systemic disease.
* Asthma- Use of inhaled corticosteroids in the last 4 weeks, use of oral steroids in the last 6 months, use of anti- inflammatory meds including statins, antihistamines, NSAIDs, salicylates, anti-rheumatics, use of any OTC medications, exacerbation requiring hospitalisation the last year, URTI within the last six months, significant CVS or inflammatory disease.
* IPF- Use of anti- inflammatory meds including statins, antihistamines, NSAIDs, salicylates, anti-rheumatics, use of oral steroids for 6 months, use of anti-fibrotic therapy( pirfendidone, nintedanib) for 6 months, FVC < 50%, baseline spO2 < 90%, use of any OTC medications, URTI within the last 6 weeks, significant CVS disease.
* Sarcoidosis- Same as IPF, including use of methotrexate for 6 months.
* COPD- Same as asthma volunteers and includes atopy.
* TB- Same as IPF, including use of anti-TB drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population include the following patients:
  Idiopathic Pulmonary fibrosis, asthma, Chronic obstructive pulmonary disease, tuberculosis,sarcoidosis and healthy
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of levels of inflammation, coagulation, complement activation and fibrosis in MLF | 3 years
  Determining biomarkers and molecular signatures(combination of mediators) in terms of cytokines and chemokines, coagulation, complement activation and fibrosis in the MLF from a range of lung diseases. The panel of mediators we aim to measure are as follows:
  Type 2 inflammation, IL-1 family and vascular injury

SECONDARY OUTCOMES:
Transcriptomics on upper and lower airway cell samples | 3 years
  These samples can then be used for the analysis of cells by flow cytometry and to determine mRNA expression(transcriptomics). The following samples will be used for cell sampling:
  Nasal curettage, bronchial and tracheal cell sampling and Mediastinal lymph node sampling(EBUS only). Several patients who have respiratory diseases such as tuberculosis and sarcoidosis have enlargement of their mediastinal lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Onn Min Kon, MBBS,MRCP,FRCP, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College NHS trust , St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No